CLINICAL TRIAL: NCT01399736
Title: Fractional Flow Reserve Guided Primary Multivessel Percutaneous Coronary Intervention to Improve Guideline Indexed Actual Standard of Care for Treatment of ST-elevation Myocardial Infarction in Patients With Multivessel Coronary Disease
Brief Title: Comparison Between FFR Guided Revascularization Versus Conventional Strategy in Acute STEMI Patients With MVD.
Acronym: CompareAcute
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maasstad Hospital (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Compare-Acute
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-05

CONDITIONS: Myocardial Infarction; Multivessel Coronary Artery Disease
Keywords: PCI FFR STEMI MVD; FFR guided PCI in acute STEMI patients with MVD
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FFR-guided revascularisation strategy (Active Comparator): In the FFR-group all flow limiting (FFR≤0.80) lesions will receive treatment by PCI and stenting. The non-IRA PCI should be performed during the same intervention. Exceptions can be made for complex lesions where the operator estimates that the revascularisation procedure will require significant contrast overload which may lead to deterioration of cardiac and renal function of the patient. Such procedures can be performed in a second procedure which should take place within the same hospitalisation. All lesions with a FFR measurement of >0.80 will not be treated.
  Interventions: Procedure: FFR-guided revascularisation strategy
- randomised to guidelines group (Placebo Comparator): In the randomised to guidelines group the procedure will stop after the FFR measurements and the patient will be referred to his treating cardiologist who will decide whether a staged PCI of the non-IRA artery should take place. The treating cardiologist will be blinded for the FFR measurements (but not angiographic imaging) and must make a decision based on conventional non-invasive ischemia detecting tests or clinical signs and symptoms i.e. very typical angina symptoms in patients with angiographic significant stenosis).
  Interventions: Procedure: randomised to guidelines group

INTERVENTIONS:
Procedure: FFR-guided revascularisation strategy — FFR-guided revascularisation strategy
  Arms: FFR-guided revascularisation strategy
Procedure: randomised to guidelines group — Staged revascularisation by proven ischemia or persistence of symptoms of angina
  Arms: randomised to guidelines group

SUMMARY:
The Compare-Acute trial is a prospective randomised trial in patients with multivessel disease, who are admitted into hospital with a ST-elevation Myocardial Infarction. The purpose of the study is to compare a FFR guided multivessel PCI taking place during the primary PCI with a primary PCI of the culprit vessel only.

Patients will be enrolled after successful revascularisation of the culprit vessel. Patients that have at least one lesion with a diameter of stenosis of more than 50% on visual estimation, feasible (operators judgement) for treatment with PCI in a non-infarct related artery, will be randomised either to the FFR guided complete revascularisation arm or staged revascularisation by proven ischemia or persistence of symptoms of angina.

Approximately 885 patients will be entered in the study.

Study hypothesis: FFR-guided complete percutaneous revascularisation of all flow-limiting stenoses in the non-IRA performed within the same procedure as the primary PCI or within the same hospitalisation will improve clinical outcomes compared to the staged revascularisation, guided by prove of ischemia or clinical judgment, as recommended from the guidelines.

DETAILED DESCRIPTION:
Background of the study: At the moment the general opinion is divided over the way the non culprit lesions in patients presenting with STEMI should be treated. While the previous guidelines stead that these lesions should be treated in a second time ( ie not during the primary intervention) the actual guidelines do not touch this argument. The reason is that the studies where the previous guidelines were based are old. Meanwhile small sized randomised trials from EU region have proven favourable outcomes with NON infarct related artery during the primary procedure while registers (non randomised trials) from USA still recommend the staged treatment. For this reason we have decided to perform a randomised study to address this issue incorporating the state of the art diagnosis and treatment, as well as the new medical therapy and PCI techniques.

Objective of the study: FFR-guided complete percutaneous revascularisation of all flow-limiting stenoses in the non-IRA performed within the same procedure as the primary PCI or within the same hospitalisation will improve clinical outcomes compared to the staged revascularisation, guided by prove of ischemia or clinical judgment, as recommended from the guidelines

Study design: Prospective, 1: 2 randomisation. FFR guided revascularisation during primary PCI (1) versus following actual guidelines (2)

Study population: All STEMI patients between 18-85 years who will be treated with primary PCI in < 12 h (more than 12 hr if persisting pain allowed) after the onset of symptoms and have at least one stenosis of >50% in a non-IRA judged feasible for treatment with PCI.

Intervention (if applicable): FFR-guided complete percutaneous revascularisation of all flow-limiting stenoses in the non-IRA performed within the same procedure as the primary PCI or within the same hospitalisation will improve clinical outcomes compared to the staged revascularisation, guided by prove of ischemia or clinical judgment, as recommended from the guidelines

Primary study parameters/outcome of the study: Composite endpoint of all cause mortality non-fatal Myocardial Infarction, any Revascularisation and Stroke (MACCE) at 12 months

ELIGIBILITY:
Inclusion Criteria:

* All patients between 18-85 years presenting with STEMI who will be treated with primary PCI in < 12 h after the onset of symptoms* and have at least one stenosis of >50% in a non-IRA on QCA or visual estimation of baseline angiography and judged feasible for treatment with PCI by the operator.

  * Patients with symptoms for more than 12 hr but ongoing angina complaints can be randomised

Exclusion Criteria:

1. Left main stem disease (stenosis > 50%)
2. STEMI due to in-stent thrombosis
3. Chronic total occlusion of a non-IRA
4. Severe stenosis with TIMI flow ≤ II of the non-IRA artery.
5. Non-IRA stenosis not amenable for PCI treatment (operators decision)
6. Complicated IRA treatment, with one or more of the following;

   * Extravasation,
   * Permanent no re-flow after IRA treatment (TIMI flow 0-1),
   * Inability to implant a stent
7. Known severe cardiac valve dysfunction that will require surgery in the follow-up period.
8. Killip class III or IV already at presentation or at the completion of culprit lesion treatment.
9. Life expectancy of < 2 years.
10. Intolerance to Aspirin, Clopidogrel, Prasugrel, Ticagrelor, Heparin, Bivaluridin, or Everolimus and known true anaphylaxis to prior contrast media of bleeding diathesis or known coagulopathy.
11. Gastrointestinal or genitourinary bleeding within the prior 3 months,
12. Planned elective surgical procedure necessitating interruption of thienopyridines during the first 6 months post enrolment.
13. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
14. Pregnancy or planning to become pregnant any time after enrolment into this study.
15. Inability to obtain informed consent.
16. Expected lost to follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 885 (Actual)
Dates: Start 2011-07; Primary Completion 2016-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Smits, MD. PHD, Principal Investigator — Maastadhospital / MCR; Elmir Omerovic, MD PhD, Study Chair — Sahlgrenska Hospital Götheborg; Gert Richardt, MD PhD, Study Chair — Herzzentrum Segeberger Kliniken; Franz-Josef Neumann, MD PhD, Study Chair — Herz-Zentrum Bad Krozingen
Locations (26):
- Czechia (3):
  - University Hospital BRNO, Brno
  - University Hospital Hradec Králové, Hradec Králové
  - Liberec Regional Hospital, Liberec
- Germany (5):
  - Herz-Zentrum Bad Krozingen, Bad Krozingen
  - Herzzentrum Bad Segeberger Klinik, Bad Segeberg
  - Klinikum Links der Weser, Bremen
  - Medizinische Klinik IV, Ingolstadt
  - Medical University Rostock, Rostock
- Hungary (4):
  - Gottsegen György Országos Kardiológiai Intézet, Budapest
  - Szabolcs - Szatmár - Bereg County Hospitals and University Teaching Hospital, Nyíregyháza
  - Szent-Györgyi Albert Klinika, Szeged
  - Zala Megyei Korhaz, Zalaegerszeg
- Netherlands (6):
  - Rijnstate Hospital, Arnhem
  - University Medical Center Groningen, Groningen
  - Atrium MC Parkstad, Heerlen
  - Maastricht Universitair Medical center, Maastricht
  - Maasstadhospital, Rotterdam
  - Medisch Centrum Haaglanden, The Hague
- Oslo University Hospital, Oslo, Norway
- Poland (4):
  - Miedziowe Centrum Zdrowia Lubin, Lubin
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
  - Kliniki Kardiologii Allenort, Warsaw
  - 4 Wojskowy Szpital Kliniczny z Polikliniką SP ZOZ, Wroclaw
- Singapore (2):
  - Tan Tock Seng Hospital, Singapore
  - Khoo Teck Puat Hospital, Singapore
- Sahlgrenska Götheborg University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piroth Z, Fulop G, Boxma-de Klerk BM, Abdelghani M, Omerovic E, Andreka P, Fontos G, Neumann FJ, Richardt G, Smits PC. Correlation and Relative Prognostic Value of Fractional Flow Reserve and Pd/Pa of Nonculprit Lesions in ST-Segment-Elevation Myocardial Infarction. Circ Cardiovasc Interv. 2022 Feb;15(2):e010796. doi: 10.1161/CIRCINTERVENTIONS.121.010796. Epub 2022 Jan 20. PMID 35045732
- [Derived] Wang LJ, Han S, Zhang XH, Jin YZ. Fractional flow reserve-guided complete revascularization versus culprit-only revascularization in acute ST-segment elevation myocardial infarction and multi-vessel disease patients: a meta-analysis and systematic review. BMC Cardiovasc Disord. 2019 Mar 1;19(1):49. doi: 10.1186/s12872-019-1022-6. PMID 30823897
- [Derived] Smits PC, Abdel-Wahab M, Neumann FJ, Boxma-de Klerk BM, Lunde K, Schotborgh CE, Piroth Z, Horak D, Wlodarczak A, Ong PJ, Hambrecht R, Angeras O, Richardt G, Omerovic E; Compare-Acute Investigators. Fractional Flow Reserve-Guided Multivessel Angioplasty in Myocardial Infarction. N Engl J Med. 2017 Mar 30;376(13):1234-1244. doi: 10.1056/NEJMoa1701067. Epub 2017 Mar 18. PMID 28317428

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Started | 295 | 590
Completed | 291 | 586
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: 885 patients with STEMI and multivessel disease
Groups:
- Total: Total of all reporting groups
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group | Total
Number analyzed (Participants) | 295 | 590 | 885
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (10) | 61 (10) | 62 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 140 | 202
  Male | 233 | 450 | 683
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Collection of race has been done, but only specified as white race and other Population: information missing for 1 patient
  Participants
    white race: number analyzed (Participants) | 295 | 589 | 884
    white race | 263 | 545 | 808
    other races | 32 | 44 | 76
BMI [Median (Full Range); unit: kg/m^2] | 27.2 [18.0 to 44.1] | 27.1 [17.7 to 54.3] | 27.1 [17.7 to 54.3]
Diabetes Mellitus [Count of Participants; unit: Participants] | 43 | 94 | 137
Hypertension [Count of Participants; unit: Participants] | 136 | 282 | 418
current smoker [Count of Participants; unit: Participants] — Population: information about smoking missing for few patients
  Participants
    number analyzed (Participants) | 294 | 589 | 883
    (all) | 120 | 287 | 407
Hypercholesterolemia [Count of Participants; unit: Participants] | 95 | 176 | 271
Family history of premature coronary artery disease [Count of Participants; unit: Participants] — Population: information missing for 1 patient
  Participants
    number analyzed (Participants) | 294 | 590 | 884
    (all) | 103 | 223 | 326
Previous stroke [Count of Participants; unit: Participants] | 10 | 26 | 36
Previous Myocardial Infarction [Count of Participants; unit: Participants] | 22 | 48 | 70
Previous PCI [Count of Participants; unit: Participants] | 25 | 44 | 69
Renal Impairment [Count of Participants; unit: Participants] | 3 | 7 | 10
Peripheral vessel disease [Count of Participants; unit: Participants] | 10 | 23 | 33
Location of infarct - Posterior [Count of Participants; unit: Participants] | 53 | 96 | 149
Location of infarct - Anterior [Count of Participants; unit: Participants] | 105 | 206 | 311
Location of infarct - Inferior [Count of Participants; unit: Participants] | 149 | 307 | 456
Location of infarct - Lateral [Count of Participants; unit: Participants] | 41 | 86 | 127
Location of infarct - impossible to determine [Count of Participants; unit: Participants] | 3 | 4 | 7
Time from symptom onset to primary PCI < 6 hr [Count of Participants; unit: Participants] | 225 | 462 | 687
Time from symptom onset to primary PCI 6-12 hr [Count of Participants; unit: Participants] | 47 | 84 | 131
Time from symptom onset to primary PCI >12 hr [Count of Participants; unit: Participants] | 23 | 44 | 67
Nr. of arteries with stenosis 2 [Count of Participants; unit: Participants] | 204 | 396 | 600
Nr. of arteries with stenosis 3 [Count of Participants; unit: Participants] | 91 | 194 | 285
Killip class >=2 [Count of Participants; unit: Participants] | 15 | 30 | 45
Maximum creatinine kinase level [Median (Full Range); unit: IU/liter] | 1040 [102 to 8182] | 1125 [112 to 11052] | 1083 [102 to 11052]
Mean time for index procedure - min [Mean (Standard Deviation); unit: minutes] | 65 (31) | 59 (28) | 61 (29)
Mean volume of contract used during index PCI [Mean (Standard Deviation); unit: ml] | 224 (104) | 202 (75) | 209 (86)
FFR procedure successful [Count of Participants; unit: Participants] | 292 | 575 | 867
Patients with lesions FFR<=0.80 [Count of Participants; unit: Participants] — Population: FFR not performed in all patients
  Participants
    number analyzed (Participants) | 292 | 575 | 867
    (all) | 158 | 275 | 433
Patients with lesions FFR>0.80 [Count of Participants; unit: Participants] — Population: FFR not performed in all patients
  Participants
    number analyzed (Participants) | 292 | 575 | 867
    (all) | 134 | 300 | 434
Mean FFR value [Mean (Standard Deviation); unit: Ratio] — Population: FFR not performed in all patients
  Ratio
    number analyzed (Participants) | 292 | 590 | 882
    (all) | 0.78 (0.12) | 0.79 (0.12) | 0.78 (0.12)
Patients with treated (FFR-guided) non-IRA lesions [Count of Participants; unit: Participants] | 163 | 0 | 163
Patients with treated (FFR-guided) non-IRA lesions during index PCI [Count of Participants; unit: Participants] | 136 | 0 | 136
Patients with treated (FFR-guided) non-IRA lesions delayed during index hospitalization [Count of Participants; unit: Participants] | 27 | 0 | 27
Patients with treated (FFR-guided) non-IRA lesions - DES only [Count of Participants; unit: Participants] | 161 | 0 | 161
Patients with treated (FFR-guided) non-IRA lesions - bare metal stent only [Count of Participants; unit: Participants] | 1 | 0 | 1
Patients with treated (FFR-guided) non-IRA lesions - balloon dilatation only [Count of Participants; unit: Participants] | 1 | 0 | 1
Patients with treated (FFR-guided) non-IRA lesions - mean nr. of stents used per patient [Mean (Standard Deviation); unit: mm] | 1.6 (0.9) | 0 (0) | 1.6 (0.9)
Patients with treated (FFR-guided) non-IRA lesions -mean length of stent [Mean (Standard Deviation); unit: mm] | 34.3 (21.0) | 0 (0) | 34.3 (21.0)
Patients with treated (FFR-guided) non-IRA lesions - mean diameter of stent [Mean (Standard Deviation); unit: mm] | 2.9 (0.4) | 0 (0) | 2.9 (0.4)
length of hospital stay [Median (Full Range); unit: days] | 4 [1 to 35] | 4 [1 to 71] | 4 [1 to 71]
Patients receiving predischarge noninvasive stress tests [Count of Participants; unit: Participants] | 21 | 71 | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Composite Endpoint of MACCE
Description: Number of participants with the composite endpoint of all cause mortality non-fatal Myocardial Infarction, any Revascularisation and Cerebrovascular Events (MACCE) at 12 months between groups
Time Frame: 12 months
Population: Patients with STEMI and multivessel disease
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 23 | 121
Statistical Analysis 1: Comparison: FFR-guided Revascularisation Strategy vs Randomised to Guidelines Group; Test type: Superiority; p < 0.001, Chi-squared; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.22 to 0.55]

2. Primary Outcome: Number of Participants With Death From Any Cause
Description: Number of participants with all cause mortality at 12 months between groups
Time Frame: 12 months
Population: Patients with STEMI and multivessel disease
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 4 | 10
Statistical Analysis 1: Comparison: FFR-guided Revascularisation Strategy vs Randomised to Guidelines Group; Test type: Superiority; p = 0.70, Chi-squared; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.25 to 2.56]

3. Primary Outcome: Number of Participants With Cardiac Death
Description: Number of participants with Cardiac mortality at 12 months between groups
Time Frame: 12 months
Population: Patients with STEMI and multivessel disease
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 3 | 6
Statistical Analysis 1: Comparison: FFR-guided Revascularisation Strategy vs Randomised to Guidelines Group; Test type: Superiority; p = 1.00, Chi-squared; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.25 to 4.01]

4. Primary Outcome: Number of Participants With Spontaneous MI
Description: Number of participants with Spontaneous Myocardial Infarction at 12 months between groups
Time Frame: 12 months
Population: Patients with STEMI and multivessel disease
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 5 | 17
Statistical Analysis 1: Comparison: FFR-guided Revascularisation Strategy vs Randomised to Guidelines Group; Test type: Superiority; p = 0.10, Chi-squared; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.22 to 1.13]

5. Primary Outcome: Number of Participants With Periprocedural MI
Description: Number of participants with Periprocedural Myocardial Infarction at 12 months between groups
Time Frame: 12 months
Population: Patients with STEMI and multivessel disease
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 2 | 11
Statistical Analysis 1: Comparison: FFR-guided Revascularisation Strategy vs Randomised to Guidelines Group; Test type: Superiority; p = 0.29, Chi-squared; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.22 to 1.59]

6. Primary Outcome: Number of Participants With Revascularization - PCI
Description: Number of participants with revascularization PCI at 12 months between groups
Time Frame: 12 months
Population: Patients with STEMI and multivessel disease
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 15 | 98
Statistical Analysis 1: Comparison: FFR-guided Revascularisation Strategy vs Randomised to Guidelines Group; Test type: Superiority; p < 0.001, Chi-squared; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.24 to 0.57]

7. Primary Outcome: Number of Participants With Revascularization - CABG
Description: Number of participants with revascularization CABG at 12 months between groups
Time Frame: 12 months
Population: Patients with STEMI and multivessel disease
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 3 | 5
Statistical Analysis 1: Comparison: FFR-guided Revascularisation Strategy vs Randomised to Guidelines Group; Test type: Superiority; p = 0.80, Chi-squared; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.29 to 5.02]

8. Primary Outcome: Number of Participants With Cerebrovascular Event
Description: Number of participants with Cerebrovascular event at 12 months between groups
Time Frame: 12 months
Population: Patients with STEMI and multivessel disease
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 0 | 4

9. Secondary Outcome: Number of Participants With Composite Endpoint of NACE (Any First Event)
Description: Number of participants with Composite endpoint of Cardiac death, Myocardial Infarction, any Revascularisation, Stroke and Major bleeding at 12 months (NACE i.e. Net Adverse Clinical Events)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 25 | 174

10. Secondary Outcome: Number of Participants With Death From Any Cause or MI
Description: Number of participants with Part of composite NACE-Death from any cause or Myocardial Infarction at 12 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 11 | 38

11. Secondary Outcome: Number of Participants With Major Bleeding
Description: Number of participants with Major bleeding at 12 months - Part of composite NACE
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 3 | 8

12. Secondary Outcome: Number of Participants With Any Bleeding at 12 Months
Description: Number of participants with any bleeding at 12 months - part of composite endpoint NACE
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 9 | 28

13. Secondary Outcome: Number of Participants With Any Bleeding at 48 Hours
Description: Number of participants with any bleeding at 48 hours - part of composite endpoint NACE
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 5 | 8

14. Secondary Outcome: Number of Participants With Hospitalization
Description: Number of participants with hospitalization for heart failure, unstable angina or chest pain
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 13 | 47

15. Secondary Outcome: Number of Participants With Revascularization
Description: Number of participants with any revascularization-Part of composite endpoint NACE
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 19 | 161

16. Secondary Outcome: Number of Participants With Stent Thrombosis
Description: Number of participants with Stent Thrombosis - Part of composite endpoint NACE
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 2 | 1

17. Secondary Outcome: Number of Participants With Primary Endpoint Outcome MACCE (Any First Event) at 3 Year
Description: Number of participants with Composite primary endpoint MACCE (any first event) at 3 year
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 46 | 178

18. Secondary Outcome: Number of Participants With All Cause Death at 3 Year
Description: Number of participants with Composite endpoint MACCE (any first event) at 3 year - all cause death
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 9 | 21

19. Secondary Outcome: Number of Participants With Cardiac Death at 3 Year
Description: Number of participants with Composite endpoint MACCE (any first event) at 3 year - Cardiac death
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 5 | 8

20. Secondary Outcome: Number of Participants With Spontaneous MI at 3 Year
Description: Number of participants with Composite endpoint MACCE (any first event) at 3 year - Spontaneous MI
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 17 | 40

21. Secondary Outcome: Number of Participants With Peri-procedural MI at 3 Year
Description: Number of participants with Composite endpoint MACCE (any first event) at 3 year - Peri-procedural MI
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 3 | 13

22. Secondary Outcome: Number of Participants With Urgent Revascularization at 3 Year
Description: Number of participants with Composite endpoint MACCE (any first event) at 3 year - urgent revascularisation
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 22 | 85

23. Secondary Outcome: Number of Participants With Elective Revascularization at 3 Year
Description: Number of participants with Composite endpoint MACCE (any first event) at 3 year -elective revascularisation
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 15 | 64

24. Secondary Outcome: Number of Participants With Cerebrovascular Event
Description: Number of participants with Composite endpoint MACCE (any first event) at 3 year -Cerebrovascular event
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 1 | 7

25. Secondary Outcome: Number of Participants With Composite Endpoint of NACE (Any First Event) at 3 Year
Description: Number of participants with Composite endpoint of Cardiac death, Myocardial Infarction, any Revascularisation, Stroke and Major bleeding at 3 year (NACE i.e. Net Adverse Clinical Events)
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 45 | 215

26. Secondary Outcome: Number of Participants With Death From Any Cause or MI
Description: Number of participants with Part of composite NACE-Death from any cause or Myocardial Infarction at 3 year
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 28 | 73

27. Secondary Outcome: Number of Participants With Major Bleeding at 3 Year
Description: Number of participants with Part of composite endpoint NACE- Major bleeding at 3 year
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 3 | 8

28. Secondary Outcome: Number of Participants With Hospitalization
Description: Number of participants with Hospitalization for heart failure, unstable angina, MI
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 28 | 75

29. Secondary Outcome: Number of Participants With Hospitalization at 3 Year
Description: Number of participants with Hospitalization for heart failure, unstable angina, MI and/or chest pain
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 30 | 87

30. Secondary Outcome: Number of Participants With Stent Thrombosis at 3 Year
Description: Number of participants with Stent Thrombosis at 3 year - Part of composite endpoint NACE
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 4 | 12

31. Secondary Outcome: Number of Participants With Any Bleeding at 3 Year
Description: Number of participants with any bleeding at 3 year - Part of composite endpoint NACE
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
Number analyzed (Participants) | 295 | 590
Participants | 4 | 12

32. Other Pre Specified Outcome: A Comparison of the Number of Patients in Both Groups With Treated Lesions With FFR ≤ 0.80 Versus Patients With Untreated Lesions With FFR ≤ 0.80;
Description: FFR+/PCI+ vs FFR+/PCI- Comparison of patients having FFR positive lesions that underwent revascularization during index procedure or in staged procedures within 45 days (groups A+C, n=202 patients) with patients having FFR positive lesions that did not undergo revascularization (group D, n=231 patients),
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Groups:
- FFR+ and PCI+: patients having FFR positive lesions that underwent revascularization during index procedure or in staged procedures within 45 days
- FFR+ and PCI-: patients having FFR positive lesions that did not undergo revascularization
Arm/Group | FFR+ and PCI+ | FFR+ and PCI-
Number analyzed (Participants) | 202 | 231
Participants | 35 | 90

33. Other Pre Specified Outcome: Comparison of Acute Versus Staged PCI for Lesions With FFR ≤ 0.80
Description: Comparison of acute versus staged PCI treatment for lesions with FFR
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Groups:
- Acute Treatment FFR+: Patients with acute PCI treatment for lesions with FFR ≤ 0.80
- Staged Treatement FFR+: Patients with staged PCI treatment for lesions with FFR ≤ 0.80
Arm/Group | Acute Treatment FFR+ | Staged Treatement FFR+
Number analyzed (Participants) | 155 | 44
Participants | 25 | 10

34. Other Pre Specified Outcome: Comparison of PCI vs Medical Therapy in FFR Negative Lesions
Description: comparison of patients receiving staged PCI treatment of FFR-negative lesions in the non-IRA (decision made by referring physician who was blinded to FFR results) and patients receiving medical therapy for FFR-negative lesions in the non-IRA
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Groups:
- FFR- Lesions Treated With PCI: patients receiving staged PCI treatment of FFR-negative lesions in the non-IRA (decision made by referring physician who was blinded to FFR results)
- FFR- Lesions Treated With Medical Therapy: patients receiving medical therapy for FFR-negative lesions in the non-IRA
Arm/Group | FFR- Lesions Treated With PCI | FFR- Lesions Treated With Medical Therapy
Number analyzed (Participants) | 13 | 418
Participants | 6 | 91

35. Post Hoc Outcome: Per Protocol Analysis - Occurence of MACCE at 3 Year
Description: post-hoc, per-protocol analysis, 328 underwent FFR-guided complete revascularization and 550 patients underwent IRA-only treatment, occurence of MACCE at 3 year
Time Frame: 3 year
Measure: Count of Participants; unit: Participants
Groups:
- FFR Guided Complete Revascularisation: Patients who underwent FFR guided complete revascularisation
- IRA Only Treatment: Patients who underwent IRA only treatment
Arm/Group | FFR Guided Complete Revascularisation | IRA Only Treatment
Number analyzed (Participants) | 328 | 550
Participants | 55 | 168

ADVERSE EVENTS:
Time Frame: 3 year
Arm/Group | FFR-guided Revascularisation Strategy | Randomised to Guidelines Group
All-Cause Mortality (participants affected / at risk) | 9/295 | 21/590
Serious Adverse Events (participants affected / at risk) | 92/295 | 308/590
Other Adverse Events (participants affected / at risk) | 12/295 | 32/590
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FFR-guided Revascularisation Strategy (N=295) | Randomised to Guidelines Group (N=590)
Myocardial Infarction (Cardiac disorders) | 20 (20) | 53 (53)
PCI (Cardiac disorders) | 34 (34) | 144 (144)
Coronary Artery Bypass graft (Cardiac disorders) | 3 (3) | 5 (5)
Cerebrovascular event (Vascular disorders) | 1 (1) | 7 (7)
Stent Thrombosis (Cardiac disorders) | 4 (4) | 12 (12)
Cardiac Hospitalisations (Cardiac disorders) | 30 (30) | 87 (87)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FFR-guided Revascularisation Strategy (N=295) | Randomised to Guidelines Group (N=590)
any bleeding (Blood and lymphatic system disorders) | 12 (12) | 32 (32) — any bleeding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT01399736/Prot_SAP_000.pdf